CLINICAL TRIAL: NCT04854096
Title: A Phase 2b, Open-label, Multicenter, Randomized, Controlled, 2-Arm Study to Assess the Efficacy and Safety of Orally Administered NS-018 Versus Best Available Therapy in Subjects With Primary Myelofibrosis, Post Polycythemia Vera Myelofibrosis, or Post-Essential Thrombocythemia Myelofibrosis With Severe Thrombocytopenia (Platelet Count <50,000/μL)
Brief Title: Study to Assess Efficacy and Safety of NS-018 Compared to BAT in Patients With Myelofibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to a business decision.
Sponsor: NS Pharma, Inc. (Industry)
Collaborators: Nippon Shinyaku Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NS-018-201
Record Dates: First submitted 2021-04-09; First posted 2021-04-22 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Primary Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis; Post-polycythemia Vera Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NS-018 (Experimental): Self-administered NS-018 300 mg orally, twice daily, preferably at the same time each day in consecutive 4-week (28-day) cycles
  Interventions: Drug: NS-018
- Best Available Therapy (BAT) (Active Comparator): Single agent per Investigator discretion or no therapy
  Interventions: Drug: Best Available Therapy

INTERVENTIONS:
Drug: NS-018 — Experimental
  Arms: NS-018
Drug: Best Available Therapy — Active Comparator
  Arms: Best Available Therapy (BAT)

SUMMARY:
This study will enroll male and female subjects who are 18 years of age or older with Primary Myelofibrosis, post-polycythemia Vera Myelofibrosis, or post-essential Thrombocythemia Myelofibrosis with severe thrombocytopenia (platelet count <50,000/µL) including subjects with intermediate-2 or high-risk MF according to the Dynamic International Prognostic Scoring System (DIPSS).

DETAILED DESCRIPTION:
NS-018 will be self-administered orally at a dose of 300 mg BID. The BAT will be administered according to manufacturer's instructions and Investigator discretion. Subjects will complete study visits at Screening, Day 1 and Day 15 of Cycle 1, 2, 3, 4, 5, 6 and Day 1 of every cycle thereafter. At these visits, blood/urine sampling, spleen measurements, bone marrow assessments, patient-reported outcome (PRO) assessments, and safety assessments may be performed.

ELIGIBILITY:
Inclusion Criteria:

* Primary MF, post-PVMF or post-ETMF according to the DIPSS risk categories of intermediate-2 or high-risk MF
* Average platelet count of <50,000/µL at Screening based on 2 measurements taken on different days; both measurements must be <50,000/µL.
* ECOG performance status ≤2.
* Life expectancy >6 months.
* Spleen volume of at least 450 cm3 measured by MRI (or by CT for applicable subjects).
* Total Symptom Score (TSS) ≥10 on the Myelofibrosis Symptom Assessment Form (MFSAF) version 4.0.
* Peripheral blast count <10%.
* No MF-directed treatment for at least 2 weeks prior to initiation of NS-018, including JAK inhibitor, erythropoietic, thrombopoietic agent, or any use of corticosteroids for MF symptom or blood count management. Low dose corticosteroids <10 mg/day prednisone or equivalent is allowed for non-MF purposes.

Exclusion Criteria:

* Active, uncontrolled systemic infection.
* Any prior treatment with more than two JAK inhibitors.
* Previous treatment with NS-018.
* Subjects actively receiving a concurrent investigational agent.
* Subjects with any unresolved AE greater than Grade 1 other than hematological AEs from previous anticancer therapy.
* Currently taking medication that is substantially metabolized by cytochrome P450 (CYP) 1A2 or CYP3A4 (see Appendix 5) or taking medication known to be strong inhibitors or inducers of CYP3A4 (see Appendix 5).
* Radiation therapy for splenomegaly within 6 months prior to study entry (screening).
* History of splenectomy or planning to undergo splenectomy.
* Subjects with a serious cardiac condition within the past 6 months such as uncontrolled arrhythmias, myocardial infarction, angina or heart disease
* Subjects diagnosed with another malignancy within 2 years prior to an enrollment.
* Subjects who have had surgery (other than placement of vascular access and bone marrow biopsy) within 4 weeks of study entry (screening), or subjects with incomplete recovery from any prior surgical procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (51):
- United States (3):
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Houston Methodist Hospital, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
- Germany (4):
  - Hamatologisch-onkologische Praxis Heinric/Bangerter Ausgsburg GbR, Augsburg
  - Universitaetsklinikum Halle (Saale), Halle
  - Universitaetsklinikum Jena, Jena
  - Universitätsmedizin Rostock, Rostock
- Italy (15):
  - AO SS Antonio, Alessandria
  - Azienda Ospedaliera SS. Antonio, Alessandria
  - ASST Spedali Civili di Brescia, Brescia
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
  - AOU "Policlinico - San Marco", Catania
  - ASST Fatebenefratelli Sacco, Milan
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - AO di Rilievo Ntl A Cardarelli, Naples
  - Azienda Ospedaliera di Rilievo Nazionale, Naples
  - AO di Rilievo Nazionale, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Istituto Nazionale Tumori Regina Elena IRCCS, Roma
  - Azienda Ospedaliera Universitaria Policlinico Umberto I, Roma
  - AO Uni Policlinico Umberto I, Rome
- Malaysia (8):
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Ampang, Ampang
  - Hospital Sultanah Aminah, Johor Bahru
  - Hospital Raja Perempuan Zainab II, Kota Bharu
  - Hospital Queen Elizabeth, Kota Kinabalu
  - University Malaya Medical Centre, Kuala Lumpur
  - Sunway Medical Centre, Petaling Jaya
  - Hospital Pulau Pinang, Pulau Pinang
- Poland (3):
  - Szpital Uniwersytecki nr 2 im. dr J. Biziela, Bydgoszcz
  - Pratia Onkologia Katowice, Katowice
  - Dolnośląskie Centrum Onkologii we Wrocławiu, Oddział Hematologiczny, Wroclaw
- South Korea (5):
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Banpo-dong
  - Gachon University Gil Medical Center, Incheon
  - Gyeongsang National University Hospital, Jinju
  - CHA Bundang Medical Center, CHA University, Seongnam
  - Soon Chun Hyang Central Medical Center, Seoul
- Thailand (2):
  - Srinagarind Hospital, Khon Kaen
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (4):
  - Istanbul Medipol University, Bağcılar, Istanbul
  - Ege Universitesi Tip Fak,, Izmir
  - Namik Kemal University Medicine School, Tekirdağ
  - Karadeniz Teknik Universitesi Tip Fak,, Trabzon
- United Kingdom (7):
  - Royal United Hospitals - Bath, Bath, England
  - Guys Hospital, London, England
  - University College London Hospitals, London, England
  - The Christie NHS Foundation Trust, Manchester, England
  - Derriford Hospital, Plymouth, England
  - Sandwell & West Birmingham Hospital, West Bromwich, England
  - Western General Hospital, Edinburgh, Scotland

IPD SHARING:
Plan to Share IPD: No
Submission to the FDA

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NS-018 | Best Available Therapy (BAT)
Started | 5 | 2
Completed (Study stopped early due to business reasons.) | 0 | 0 (Study stopped early due to business reasons.)
Not Completed | 5 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Study terminated by Sponsor due to business reasons. | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other reasons | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NS-018 | Best Available Therapy (BAT) | Total
Number analyzed (Participants) | 5 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.0 (16.48) | 70.5 (0.71) | 66.6 (13.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Spleen Volume
Description: Proportion of subjects who achieve ≥35% reduction in spleen volume from baseline compared to Week 24 as measured by MRI (or by CT for applicable subjects)
Time Frame: baseline and week 24
Population: The primary outcome measure for an efficacy endpoint to compare the efficacy of NS-018 to the Best Available Therapy (BAT) was analyzed among the limited participants enrolled before the study was terminated early for business reasons.
Measure: Count of Participants; unit: Participants
Arm/Group | NS-018 | Best Available Therapy (BAT)
Number analyzed (Participants) | 5 | 2
Participants | 0 | 0

2. Primary Outcome: Change in Total Symptom Score (TSS)
Description: Proportion of subjects who achieve ≥50% reduction in total symptom score from baseline compared to Week 24 as measured by the MF-SAF v4.0
Time Frame: baseline and week 24
Population: This co-primary outcome measure for an efficacy endpoint to compare NS-018 to the Best Available Therapy (BAT) was analyzed among the limited participants enrolled before the study was terminated early for business reasons. .
Measure: Count of Participants; unit: Participants
Arm/Group | NS-018 | Best Available Therapy (BAT)
Number analyzed (Participants) | 5 | 2
Participants | 0 | 1

3. Secondary Outcome: Change in Spleen Volume
Description: Proportion of subjects in NS-018 vs BAT arm who achieve ≥35% reduction in spleen volume from baseline at any time up to Week 24 as measured by MRI (or by CT for applicable subjects)
Time Frame: from baseline to anytime before or at week 24
Population: This secondary outcome measure for an efficacy endpoint to compare the efficacy of NS-018 to the Best Available Therapy (BAT) was analyzed among the limited participants enrolled before the study was terminated early for business reasons.
Measure: Count of Participants; unit: Participants
Arm/Group | NS-018 | Best Available Therapy (BAT)
Number analyzed (Participants) | 5 | 2
Participants | 1 | 0

4. Secondary Outcome: Comparison of Treatment-emergent AEs Between NS-018 and BAT
Description: Laboratory events graded by the NCI CTCAE v5.0 will be assessed in both arms, to compare the safety profile of NS-018 versus BAT.
Time Frame: from baseline to week 24
Population: TEAE's were evaluated in the participants who received NS-018 or BAT.
Measure: Count of Participants; unit: Participants
Arm/Group | NS-018 | Best Available Therapy (BAT)
Number analyzed (Participants) | 5 | 2
Participants | 5 | 2

ADVERSE EVENTS:
Time Frame: from baseline to week 24
Arm/Group | NS-018 | Best Available Therapy (BAT)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/2
Other Adverse Events (participants affected / at risk) | 5/5 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NS-018 (N=5) | Best Available Therapy (BAT) (N=2)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NS-018 (N=5) | Best Available Therapy (BAT) (N=2)
Anaemia (Blood and lymphatic system disorders) | 4 (8) | 0 (0)
Platelet Count Decrease (Investigations) | 2 (2) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Influenza-like illness (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (3)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Arthalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Venous haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was stopped early for business reasons. Therefore the efficacy outcomes were evaluated only in the limited number of patients enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UK: The Sponsor recognizes that the PI may have a responsibility to ensure that results of scientific interest arising from the Clinical Trial are appropriately published.

Germany: Details of study and its results shall not be publicized or published in any form without prior written consent of the sponsor.

Malaysia: Institution and Investigator may publish or otherwise publicly disclose, for non-commercial purposes.

DOCUMENTS (2):
  • Study Protocol (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/96/NCT04854096/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT04854096/SAP_001.pdf